CLINICAL TRIAL: NCT05865379
Title: Efficacy and Safety of BUFY01 Versus SVS20 in the Treatment of Dry Eye Disease: a Non-inferiority Investigation
Brief Title: Efficacy and Safety of BUFY01 Versus SVS20 in the Treatment of Dry Eye Disease
Acronym: BUSTON-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TRB Chemedica International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUFY01-CT-2101
Record Dates: First submitted 2023-05-01; First posted 2023-05-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BUFY01 (Experimental): 0.18% Sodium Hyaluronate (trometamol buffer) in single-dose containers of 0.3 mL
  Interventions: Device: BUFY01 eye drops in single-dose containers
- SVS20 (Active Comparator): 0.18% Sodium Hyaluronate (phosphate buffer) in single-dose containers of 0.3 mL
  Interventions: Device: SVS20 eye drops in single-dose containers

INTERVENTIONS:
Device: BUFY01 eye drops in single-dose containers — 1 to 2 drops in each eye, as often as needed
  Arms: BUFY01
Device: SVS20 eye drops in single-dose containers — 1 to 2 drops in each eye, as often as needed
  Arms: SVS20

SUMMARY:
The goal of this interventional investigation is to compare BUFY01 with SVS20 in the treatment of patients with dry eye disease. The main questions it aims to answer are:

* Is BUFY01 non-inferior to SVS20 in terms of signs of DED?
* Is BUFY01 non-inferior to SVS20 in terms of symptoms of DED?

Participants will be asked to:

* Visit the trial site at 4 different timepoints
* Use the allocated study treatment everyday until the end of the study (during 3 months)
* Be examined by the investigator
* Complete several questionnaires
* Return unused study treatment.

Researchers will compare BUFY01 to SVS20 to see if both study treatments provide similar effects on signs and symptoms of the disease, together with comparable safety.

ELIGIBILITY:
Inclusion Criteria includes:

* At least a 3-month documented history of bilateral dry eye syndrome needing artificial tears;
* At least one eye with Oxford score ≥ 4 and ≤ 9;
* At least one objective sign of tear deficiency (in at least one eligible eye);
* Having a health insurance.

Exclusion Criteria includes:

* Wear of contact lenses starting within the last 2 months;
* Best-corrected visual acuity (BCVA) < 1/10;
* Severe DED with one of the listed conditions:
* Severe blepharitis;
* Seasonal allergy;
* Any issues of the ocular surface not related to DED;
* History of ocular trauma, infection or inflammation not related to DED;
* History of ocular surgery, including laser surgery;
* Unstable glaucoma;
* Use of artificial tears with preservative within the last 2 weeks;
* Systemic (enteral or parenteral) or local (topical) use of one of the listed medications:
* Known hypersensitivity to any constituent of the study treatments;
* Pregnancy or breastfeeding;
* Participation in another clinical study within the last 90 days;
* Legally restricted autonomy, freedom of decision and action.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Signs | Day 28
  Change from baseline in Oxford score (0-15, a higher score meaning a worse outcome)

SECONDARY OUTCOMES:
Symptoms | Day 28
  Change from baseline in Ocular Surface Disease Index

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital des Quinze-Vingts, Paris
  - CHU Saint-Etienne, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No